CLINICAL TRIAL: NCT05117671
Title: Is the EBJIS Definition of Prosthetic Joint Infection Meaningful in Our Clinical Practice? - a Multicentric Validation Study
Brief Title: Is the EBJIS Definition of Prosthetic Joint Infection Meaningful in Our Clinical Practice?
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00133; mu21Clauss
Record Dates: First submitted 2021-11-10; First posted 2021-11-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Periprosthetic Joint Infection (PJI)
Keywords: Infection Likely group; Infection Unlikely group; European Bone and Joint Infection Society (EBJIS); revision total hip arthroplasty (THA); revision total knee arthroplasty (TKA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- revision total hip or knee arthroplasties: THA/TKA patients that underwent revision surgery between 01.01.2013 until 31.12.2018
  Interventions: Other: data collection to classify infection status

INTERVENTIONS:
Other: data collection to classify infection status — Review of medical records of all selected cases (TKA/THA patients) to classify infection status according to different classifications (EBJIS, MSIS/ICM 2013, ICM 2018).

SUMMARY:
This retrospective multi-center, multi-national cohort study is to validate the European Bone and Joint Infection Society (EBJIS) Definition of Prosthetic Joint Infection. Specifically, it is to analyze the outcome of the Infection Likely group and compare it to the Infection Unlikely group as well as other subgroups within previous validated definitions (Musculoskeletal Infection Society (MSIS)/International Consensus on Musculoskeletal Infection (ICM) 2013 and ICM 2018).

DETAILED DESCRIPTION:
Periprosthetic joint infection (PJI) is a major burden for healthcare systems. The European Bone and Joint Infection Society (EBJIS) proposed a new set of criteria introducing a three level 'traffic light' distinction: Infection Unlikely, Infection Confirmed but also an intermediate group called Infection Likely (but nor confirmed). This retrospective multi-center, multi-national cohort study is to validate the EBJIS Definition of Prosthetic Joint Infection. Specifically, it is to analyze the outcome of the Infection Likely group and compare it to the Infection Unlikely group as well as other subgroups within previous validated definitions (Musculoskeletal Infection Society (MSIS)/International Consensus on Musculoskeletal Infection (ICM) 2013 and ICM 2018).

ELIGIBILITY:
Inclusion Criteria:

* THA/TKA patients that underwent revision surgery regardless of final aseptic vs. infected diagnosis between 01.01.2013 until 31.12.2018

Exclusion Criteria:

* less than two years follow up
* less than four intraoperative microbiology samples (synovial fluid, tissue samples, implant sonication)
* no preoperative/intraoperative synovial fluid differential leukocyte count

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: THA/TKA patients that underwent revision surgery regardless of final aseptic vs. infected diagnosis between 1st of January 2013 until 31.12.2018. All data coming from everyday clinical work. The average patient operated with revision arthroplasty is normally aged above 70 years.
Sampling Method: Probability Sample
Enrollment: 1554 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Prosthetic Joint Infections (with or without the need for further surgery) | since 01.01.2013 with a minimum of two years follow up
  Number of Prosthetic Joint Infections (with or without the need for further surgery) among each PJI definition ("Infection Unlikely", "Infection Confirmed", "Infection Likely (but nor confirmed)"
Prosthetic Joint Infections (with or without the need for further surgery) | since 01.01.2013 with a minimum of two years follow up
  Number of Prosthetic Joint Infections (with or without the need for further surgery) according to different classifications (EBJIS, MSIS/ICM 2013, ICM 2018).
Need for Revision Surgery | since 01.01.2013 with a minimum of two years follow up
  Number of Revision Surgeries (for all causes, PJI and aseptic failure) among each PJI definition ("Infection Unlikely", "Infection Confirmed", "Infection Likely (but nor confirmed)"
Need for Revision Surgery | since 01.01.2013 with a minimum of two years follow up
  Number of Revision Surgeries (for all causes, PJI and aseptic failure) according to different classifications (EBJIS, MSIS/ICM 2013, ICM 2018).
Survival rates of different subgroups among each PJI definition | since 01.01.2013 with a minimum of two years follow up
  Survival rates of different subgroups among each PJI definition ("Infection Unlikely", "Infection Confirmed", "Infection Likely (but nor confirmed)"
Survival rates between different definitions | since 01.01.2013 with a minimum of two years follow up
  Survival rates between different classifications (EBJIS, MSIS/ICM 2013, ICM 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Jorge Gomes de Sousa, Prof. Dr. med., Principal Investigator — Centro Hospitalar Universitario do Porto, Orthopedics Department
Locations (2):
- Centro Hospitalar do Porto, Porto, Portugal, Porto, Portugal
- University Hospital Basel, Orthopedics and Traumatology, Basel, Switzerland